CLINICAL TRIAL: NCT02696239
Title: Vaginal Cuff Closure in Robotic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6297
Record Dates: First submitted 2016-02-21; First posted 2016-03-02 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2016-02

CONDITIONS: Complications of Medical Care
Keywords: vaginal cuff closure; Robotic Hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- V-lock suture (Active Comparator): V-lock absorbable Wound Closure Device, by Covidien
  Interventions: Device: V-lock suture
- Vicryl suture (Active Comparator): Vicryl suture by Ethicon
  Interventions: Device: Vicryl Suture
- Lapra-Ty II (Active Comparator): Lapra-Ty II, Absorbable Suture Clip, by Ethicon
  Interventions: Device: Lapra-Ty II

INTERVENTIONS:
Device: V-lock suture
  Arms: V-lock suture
Device: Vicryl Suture
  Arms: Vicryl suture
Device: Lapra-Ty II
  Arms: Lapra-Ty II

SUMMARY:
The purpose of this study is to evaluate the impact of implementing different types of suturing materials and techniques of vaginal cuff closure in robotic assisted laparoscopic hysterectomy on cost, operative time and post operative surgical outcomes.

DETAILED DESCRIPTION:
Robotic assisted laparoscopic surgery is the fastest growing new modality in gynecologic surgery. Surgeons are adapting it to perform both benign and oncologic gynecologic procedures. Therefore, the fastest growing robotic procedure in the united states is hysterectomy.

The literature in laparoscopic hysterectomy, both robotic and non-robotic, reports a complication of vaginal closure disruption after hysterectomy higher than with abdominal surgery. Reasons hypothesized for this phenomenon include colpotomy (vaginal incision) technique, vaginal closure technique, and types of suture. At present, no further follow up studies have been done to test some of these hypothesis. In light of the rapid adoption of this approach to hysterectomy, more data on this issue will help the physician in counseling patients regarding complications, as well as helping surgeons choose materials and techniques in their hysterectomies which will diminish the chance for this unfortunate complication, which causes pain, hospitalization and excess morbidity after the original surgery.

Additionally, a parallel development of newer suturing materials, the so-called "barbed" self-anchoring sutures, typically fabricated from monofilament materials, have been reported used in laparoscopic hysterectomies in case series. The relative contribution of theses newer materials to the rates of cuff disruption is unknown.

The protocol proposes testing the null hypothesis that different suture materials and methods of closure do not cause a significant difference in the rates of vaginal cuff disruption after robotic assisted laparoscopic total hysterectomy.

Study design is a prospective randomized controlled trial. Patients will be blindly randomized to one of the 3 closure techniques using 3 different materials. Technique and material by necessity can not be blinded to the surgeon. Otherwise, standard surgical technique will be used. Followup in 2 and 6 weeks for clinical assessment will be performed. To asses the long term of cuff disruption, a 12 month interview will be also conducted. Data points will include operative time for closure, postoperative pain at 2 and 6 weeks, postoperative pain with urination/voiding at 2 and 6 weeks, spotting, bleeding and /or frank vaginal disruption documented at 2 and 6 weeks, and pain and presence of dyspareunia at 12 months will be assessed.

Cost associated with cuff closure will be calculated by addition of OR time and material cost.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for robotic assisted laparoscopic hysterectomy

Exclusion Criteria:

* Patients who will not consent.
* Hysterectomy due to malignant conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Vaginal cuff dehiscence | 12 months
  Postoperative inspection for vaginal cuff dehiscence

SECONDARY OUTCOMES:
Complications | 6 weeks
  Post-operative vaginal bleeding, bowel or urinary dysfunction
Operative time costs | 1 year
  Measurement of operative time and determination of unit cost per surgery
Suturing material costs | 1 year
  Comparison of the amount and type of suture utilized per surgery
Operative suturing time | During surgery
  Time to complete Vaginal cuff closure
Post operative pain | 6 weeks
  Visual Analog Scale
Vaginal bleeding/ spotting | 12 months
  Presence of postoperative vaginal bleeding
Resumption of sexual activity | 12 months
  Time to resumption of intercourse
Dyspareunia | 12 months
  Assessment of Painful Intercourse

CONTACTS AND LOCATIONS:
Overall Officials: David Eisenstein, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AAGL Advancing Minimally Invasive Gynecology Worldwide. AAGL position statement: route of hysterectomy to treat benign uterine disease. J Minim Invasive Gynecol. 2011 Jan-Feb;18(1):1-3. doi: 10.1016/j.jmig.2010.10.001. Epub 2010 Nov 6. No abstract available. PMID 21059487
- [Background] Greenberg JA, Einarsson JI. The use of bidirectional barbed suture in laparoscopic myomectomy and total laparoscopic hysterectomy. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):621-3. doi: 10.1016/j.jmig.2008.06.004. Epub 2008 Jul 10. PMID 18619922
- [Background] Einarsson JI, Vellinga TT, Twijnstra AR, Chavan NR, Suzuki Y, Greenberg JA. Bidirectional barbed suture: an evaluation of safety and clinical outcomes. JSLS. 2010 Jul-Sep;14(3):381-5. doi: 10.4293/108680810X12924466007566. PMID 21333192
- [Background] Siedhoff MT, Yunker AC, Steege JF. Decreased incidence of vaginal cuff dehiscence after laparoscopic closure with bidirectional barbed suture. J Minim Invasive Gynecol. 2011 Mar-Apr;18(2):218-23. doi: 10.1016/j.jmig.2011.01.002. PMID 21354068